CLINICAL TRIAL: NCT06286241
Title: Comparison of the Complications in Multiple Myeloma Patients Who Received Autologous Stem Cell Transplantation Between in HEPA-filtered Room and Non-HEPA-filtered Room
Acronym: Step down ward
Status: Not yet recruiting | Type: Observational
Sponsor: Siriraj Hospital (Other)
Responsible Party: Principal Investigator, Chutima Kunacheewa, lecturer, Siriraj Hospital
Other Study IDs: 877/2564(IRB2)
Record Dates: First submitted 2024-02-22; First posted 2024-02-29 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Multiple Myeloma
Keywords: multiple myeloma; autologous stem cell transplantation; HEPA-filtered room; non-HEPA-filtered room
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HEPA-filtered room: multiple myeloma patients who received autologous stem cell transplantation were admitted in HEPA-filtered room
- non-HEPA-filtered room: multiple myeloma patients who received autologous stem cell transplantation were admitted in non-HEPA-filtered room

SUMMARY:
The goal of this observational study is to comparison of the complications in multiple myeloma patients who received autologous stem cell transplantation between in HEPA-filtered room and non-HEPA-filtered room. The main questions it aims to answer are:

* The incidence of febrile neutropenia, infection, and duration of hospital stay
* 2-year progression free survival Participants will be collected the data of baseline diagnosis, treatment, treatment results and complications during admission and follow-up visits from hospital medical record.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 - 65 years old
* Patients with multiple myeloma undergoing treatment with autologous stem cell transplantation and having a Hematopoietic Cell Transplantation-Specific Comorbidity Index (HCT-CI) score less than or equal to 2
* Patients must provide signed consent to participate in the research if they undergo ASCT after the study has been approved.
* If patients undergo ASCT before the study approval, retrospective data will be collected.

Exclusion Criteria:

* Patients with concomitant other types of cancer
* Patients who refuse to participate in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: multiple myeloma patients who received autologous stem cell transplantation
Sampling Method: Probability Sample
Enrollment: 344 (Estimated)
Dates: Start 2024-03-25 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-07-30 (Estimated)

PRIMARY OUTCOMES:
febrile neutropenia | during admission
  incidence of febrile neutropenia
Infection | during admission
  incidence of Infection
duration of admission | during admission
  duration of admission
progression free survival | 2 years
  duration of survival

IPD SHARING:
Plan to Share IPD: Undecided
Need a consensus from colleagues